CLINICAL TRIAL: NCT01476566
Title: Can Diagnostics and Pharmacological Prescriptions in Patients With Heart Failure be Improved? A Cluster Randomised Educational Intervention in General Practice. A Study Protocol.
Brief Title: Can Diagnostics and Pharmacological Prescriptions in Patients With Heart Failure be Improved in General Practice?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the study was terminated before study start, no researcher was attached to the study
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Arne Fetveit, associate professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KTV-3
Record Dates: First submitted 2011-11-14; First posted 2011-11-22 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
Keywords: aged; family practice
MeSH Terms: conditions — Heart Failure | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational intervention (Experimental): A multifaceted intervention has been tailored where key components are educational outreach visits (EOV) to the CME-groups, audit, and feedback. Trained GPs will conduct the EOVs during which evidence-based recommendations for diagnosis and treatment of HF will be presented.
  Interventions: Behavioral: Educational intervention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Educational intervention — Peer continuous medical education (CME) groups in general practice will be recruited to a cluster randomised educational intervention study. Participating groups will be randomised either to an intervention- or a control group. A multifaceted intervention has been tailored where key components are educational outreach visits (EOV) to the CME-groups, audit, and feedback. Trained GPs will conduct the EOVs during which evidence-based recommendations for diagnosis and treatment of HF will be presented. A software will be handed out for installation on participants' practice computers, enabling collection of diagnosis- and prescription-data. The captured data will subsequently be linked to corresponding data from the Norwegian Prescription Database (NorPD).
  Arms: Educational intervention

SUMMARY:
This study will explore the possible effect of a tailored educational intervention towards general practitioners in Norway, in order to improve the quality of treatment for heart failure in general practice.

DETAILED DESCRIPTION:
Chronic heart failure (HF) is a syndrome with a poor prognosis and with a prevalence increasing steeply by patients' age. Studies indicate that there are large potentials for improving general practitioners' diagnosis and management of HF. We have designed an educational intervention aiming at improving GPs' diagnosis and management of HF.

Peer continuous medical education (CME) groups in general practice will be recruited to a cluster randomised educational intervention study. Participating groups will be randomised either to an intervention- or a control group. A multifaceted intervention has been tailored where key components are educational outreach visits (EOV) to the CME-groups, audit, and feedback. Trained GPs will conduct the EOVs during which evidence-based recommendations for diagnosis and treatment of HF will be presented. A software will be handed out for installation on participants' practice computers, enabling collection of diagnosis- and prescription-data. The captured data will subsequently be linked to corresponding data from the Norwegian Prescription Database (NorPD). Individual feedback reports will be sent each participant in the beginning and at the end of the study. Main outcomes measure is the proportion of HF patients prescribed an ACE-inhibitor (or an angiotensine receptor blocker) and a betablocker in combination. Baseline data will provide material for a descriptive, cross sectional study. Patient related outcomes in terms of HF-hospital admissions and all cause mortality will be obtained by record linkage with NorPD and the Norwegian Patient Registry. Included in the intervention group is also a sub-study using a pop-up programme to facilitate disclosure of non-diagnosed HF patients in own practice. Finally, we plan a questionnaire study (among GPs in intervention group and their HF-patients) to get more knowledge regarding diagnostic workup, quality of care, non-pharmacological issues, and chronic care management of HF.

ELIGIBILITY:
Inclusion Criteria:

* General practitioner
* Specialist in general practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01 (Estimated); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Whether drug-treatment of heart failure will be more adherent to guidelines after an educational intervention towards general practitioners (GPs). | 1 year
  The proportion of heart failure-patients receiving treatment with an angiotensin converting enzyme inhibitor (ACE-I) or an angiotensin-2 receptor blocker (ARB) and a beta-blocker (BB) before and after an educatopnal intervention.

SECONDARY OUTCOMES:
Hospital admissions and mortality | 1 year
  Differences in heart failure-related hospital admissions and all cause mortality between intervention group and control group.